CLINICAL TRIAL: NCT03126695
Title: An Open-label, Randomized, 4-period, 4-treatment, Cross-over, Single-center, Single-dose Study to Assess the Relative Bioavailability of Ticagrelor in Different Formulations in Healthy Adult Subjects
Brief Title: A Study to Compare if the Uptake of Ticagrelor in the Body Differs When Different Tablets Are Administered
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D5136C00011
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Sickle Cell Disease
Keywords: Abnormal hemoglobin (called hemoglobin S or sickle hemoglobin) in the red blood cells; Thrombotic cardiovascular events; Acute coronary syndrome; P2Y12 platelet inhibitor; Brilinta
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait; Acute Coronary Syndrome | interventions — Excipients; Water; Ticagrelor; Tablets

STUDY DESIGN:
Intervention Model Description: A randomized cross-over design has been chosen to minimize the effects of between-subject variability and any period effects on the overall results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1 (ADBC) (Experimental): Subjects were randomized to treatment sequence ADBC:
  On Day 1, following an overnight fast of at least 10 hours, each subject will receive single dose of the treatment assigned to that treatment period.
  A =Ticagrelor granule for oral suspension equal to 90 mg. B = Ticagrelor pediatric tablets equal to 90 mg. C= Ticagrelor pediatric tablets suspended in water equal to 90 mg. D = Ticagrelor commercial IR (1 x 90 mg) tablet
  Interventions: Drug: Ticagrelor granule; Drug: Ticagrelor pediatric tablets; Drug: Ticagrelor pediatric tablets suspended in water; Drug: Ticagrelor immediate release (IR) tablets (Commercial tablet)
- Treatment Sequence 2 (BACD) (Experimental): Subjects were randomized to treatment sequence BACD:
  On Day 1, following an overnight fast of at least 10 hours, each subjects will receive single dose of the treatment assigned to that treatment period.
  A =Ticagrelor granule for oral suspension equal to 90 mg. B = Ticagrelor pediatric tablets equal to 90 mg. C= Ticagrelor pediatric tablets suspended in water equal to 90 mg. D = Ticagrelor commercial IR (1 x 90 mg) tablet
  Interventions: Drug: Ticagrelor granule; Drug: Ticagrelor pediatric tablets; Drug: Ticagrelor pediatric tablets suspended in water; Drug: Ticagrelor immediate release (IR) tablets (Commercial tablet)
- Treatment Sequence 3 (CBDA) (Experimental): Subjects were randomized to treatment sequence CBDA:
  On Day 1, following an overnight fast of at least 10 hours, each subjects will receive single dose of the treatment assigned to that treatment period.
  A =Ticagrelor granule for oral suspension equal to 90 mg. B = Ticagrelor pediatric tablets equal to 90 mg. C= Ticagrelor pediatric tablets suspended in water equal to 90 mg. D = Ticagrelor commercial IR (1 x 90 mg) tablet
  Interventions: Drug: Ticagrelor granule; Drug: Ticagrelor pediatric tablets; Drug: Ticagrelor pediatric tablets suspended in water; Drug: Ticagrelor immediate release (IR) tablets (Commercial tablet)
- Treatment Sequence 4 (DCAB) (Active Comparator): Subjects were randomized to treatment sequence DCAB:
  On Day 1, following an overnight fast of at least 10 hours, each subjects will receive single dose of the treatment assigned to that treatment period.
  A =Ticagrelor granule for oral suspension equal to 90 mg. B = Ticagrelor pediatric tablets equal to 90 mg. C= Ticagrelor pediatric tablets suspended in water equal to 90 mg. D = Ticagrelor commercial IR (1 x 90 mg) tablet
  Interventions: Drug: Ticagrelor granule; Drug: Ticagrelor pediatric tablets; Drug: Ticagrelor pediatric tablets suspended in water; Drug: Ticagrelor immediate release (IR) tablets (Commercial tablet)

INTERVENTIONS:
Drug: Ticagrelor granule — A P2Y12 receptor inhibitor provided as granule for suspension.
Drug: Ticagrelor pediatric tablets — A P2Y12 receptor inhibitor provided as pediatric tablets to be swallowed whole.
Drug: Ticagrelor pediatric tablets suspended in water — A P2Y12 receptor inhibitor provided as pediatric tablets suspended in water.
Drug: Ticagrelor immediate release (IR) tablets (Commercial tablet) — A P2Y12 platelet inhibitor indicated to reduce the rate of thrombotic cardiovascular events in patients with acute coronary syndrome (unstable angina, non-ST (S and T waves) elevation MI or ST elevation MI) and in patients with a history of MI
  Other Names: Brilinta

SUMMARY:
To evaluate the relative bioavailability of ticagrelor for the different formulations. A randomized cross-over design has been chosen to minimize the effects of between-subject variability and any period effects on the overall results.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, 4-period, 4-treatment, cross-over, single-center, single-dose study to assess the relative bioavailability of different formulations of ticagrelor in approximately 44 healthy adult subjects. Eligible subjects will be healthy male and female aged 18 to 55 years, with a body weight of 55 to 100 kg and a body mass index (BMI) of 18 to 30 kg/m2. Of the 44 randomized subjects, at least 36 evaluable subjects should be at the end of the last treatment period. Subjects will be randomized to 1 of 4 treatment sequences and will receive single oral doses of 4 different formulations of ticagrelor under fasted conditions. Subjects will fast for at least 10 hours prior to administration of Investigational Medicinal Products (IMPs). No fluids will be allowed apart from water which can be given until 1 hour prior to administration of the IMP and then from 2 hours after administration of the IMP. A meal can be given 4 hours after administration of the IMP.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study specific procedures.
2. Healthy male and female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at Screening and on each admission to the Clinical Unit, must not be lactating and if of non child-bearing potential, confirmed at Screening by fulfilling one of the following criteria:

   - Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the post-menopausal range (> 40 milli international units per milliliter (mIU/mL)). - Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation. - Childbearing potential and are sexually active must use 1 highly effective method of birth control in combination with a barrier method, from the time of IMP administration until 3 months after the last dose of IMP.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Able to understand, read and speak the German language.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the potential subject at risk because of participation in the study, or influence the results or the potential subject's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
4. Any clinically significant abnormalities in hematology, clinical chemistry, coagulation or urinalysis results at Screening or Day -1 of Treatment Period 1, as judged by the Investigator.
5. Any clinically significant abnormal findings in vital signs at Screening or Day -1 of Treatment Period 1, as judged by the Investigator.
6. Any clinically significant abnormalities on 12-lead ECG at Screening, as judged by the Investigator.
7. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (anti-HBcAb), hepatitis C antibodies (anti- HCV) and human immunodeficiency virus (HIV) antibodies.
8. Has received a new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.
9. Plasma donation within 1 month of Screening or any blood donation/loss more than 500 mL during the 3 months prior to Screening. 10. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to ticagrelor.

11. Current smokers or those who have smoked or used nicotine products within the previous 3 months.

12. Positive screen for drugs of abuse or cotinine (cotinine level above 500 ng/mL) at Screening or on each admission to the Clinical Unit or positive screen for alcohol on each admission to the Clinical Unit.

13. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.

14. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.

15. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol, as judged by the Investigator.

16. Involvement of any AstraZeneca or Clinical Unit employee or their close relatives.

17. Judgment by the Investigator that the potential subject should not participate in the study if they have any ongoing or recent (i.e., during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.

18. Consumption of poppy seeds within 7 days of first admission to the Clinical Unit.

19. History of hemophilia, von Willebrand's disease, lupus anticoagulant, or other diseases/syndromes that can either alter or increase the propensity for bleeding. 20. A personal history of vascular abnormalities including aneurysms; a personal history of severe hemorrhage, hematemesis, melena, hemoptysis, severe epistaxis, severe thrombocytopenia, intracranial hemorrhage; or rectal bleeding within 1 year prior to Screening; or history suggestive of peptic ulcer disease; or at the discretion of the Investigator.

21. History of a clinically significant non-traumatic bleed or clinically significant bleeding risk, as judged by the Investigator.

22. Use of aspirin, ibuprofen, NSAIDs, or any other drug known to increase the propensity for bleeding for 2 weeks before randomization. 23. Platelet count less than 150 x 109/L.

24. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male and female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
Enrollment: 44 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | At 0 hours (pre-dose) and post-dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  * To determine the relative bioavailability of ticagrelor granule for oral suspension and the pediatric ticagrelor tablet to the commercial ticagrelor tablet in healthy subjects.
  * To determine the relative bioavailability of ticagrelor pediatric tablet taken whole and the pediatric tablet dispersed in water to the granule for oral suspension in healthy subjects.
  * To evaluate the bioequivalence between the pediatric ticagrelor tablet taken whole and the pediatric ticagrelor tablet dispersed in water in healthy subjects.
Area under plasma concentration-time curve from zero to infinity (AUC) | At 0 hours (pre-dose) and post-dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose.
  * To determine the relative bioavailability of ticagrelor granule for oral suspension and the pediatric ticagrelor tablet to the commercial ticagrelor tablet in healthy subjects.
  * To determine the relative bioavailability of ticagrelor pediatric tablet taken whole and the pediatric tablet dispersed in water to the granule for oral suspension in healthy subjects.
  * To evaluate the bioequivalence between the pediatric ticagrelor tablet taken whole and the pediatric ticagrelor tablet dispersed in water in healthy subjects.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUC(0-t)) | At 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  To compare the pharmacokinetic (PK) profiles of ticagrelor and its active metabolite (AR-C124910XX) in healthy subjects when administered as granule for oral suspension, pediatric ticagrelor tablet, pediatric ticagrelor tablet suspended in water and commercial ticagrelor tablet.
Time to reach maximum observed plasma concentration, taken directly from the individual concentration-time curve (tmax). | At 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  To compare the PK profiles of ticagrelor and its active metabolite (AR-C124910XX) in healthy subjects when administered as granule for oral suspension, pediatric ticagrelor tablet, pediatric ticagrelor tablet suspended in water and commercial ticagrelor tablet.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz). | At 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  To compare the PK profiles of ticagrelor and its active metabolite (AR-C124910XX) in healthy subjects when administered as granule for oral suspension, pediatric ticagrelor tablet, pediatric ticagrelor tablet suspended in water and commercial ticagrelor tablet.
Terminal rate constant, estimated by log-linear regression of the terminal part of the concentration-time curve (λz). | At 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  To compare the PK profiles of ticagrelor and its active metabolite (AR-C124910XX) in healthy subjects when administered as granule for oral suspension, pediatric ticagrelor tablet, pediatric ticagrelor tablet suspended in water and commercial ticagrelor tablet.
Apparent clearance, estimated as dose divided by AUC (ticagrelor only) (CL/F). | At 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  To compare the PK profiles of ticagrelor and its active metabolite (AR-C124910XX) in healthy subjects when administered as granule for oral suspension, pediatric ticagrelor tablet, pediatric ticagrelor tablet suspended in water and commercial ticagrelor tablet.
Apparent volume of distribution at the terminal phase, estimated by dividing the apparent clearance (CL/F) by λz (ticagrelor only) (Vz/F). | At 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  To compare the PK profiles of ticagrelor and its active metabolite (AR-C124910XX) in healthy subjects when administered as granule for oral suspension, pediatric ticagrelor tablet, pediatric ticagrelor tablet suspended in water and commercial ticagrelor tablet.
Ratio of metabolite Cmax to parent Cmax, adjusted for differences in molecular weights (MRCmax). | At 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  To compare the PK profiles of ticagrelor and its active metabolite (AR-C124910XX) in healthy subjects when administered as granule for oral suspension, pediatric ticagrelor tablet, pediatric ticagrelor tablet suspended in water and commercial ticagrelor tablet.
Ratio of metabolite AUC(0-t) to parent AUC(0-t), adjusted for differences in molecular weights (MRAUC(0-t)). | At 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  To compare the PK profiles of ticagrelor and its active metabolite (AR-C124910XX) in healthy subjects when administered as granule for oral suspension, pediatric ticagrelor tablet, pediatric ticagrelor tablet suspended in water and commercial ticagrelor tablet.
Ratio of metabolite AUC to parent AUC, adjusted for differences in molecular weights (MRAUC) | At 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose in each treatment period
  To compare the PK profiles of ticagrelor and its active metabolite (AR-C124910XX) in healthy subjects when administered as granule for oral suspension, pediatric ticagrelor tablet, pediatric ticagrelor tablet suspended in water and commercial ticagrelor tablet.
Number of patients with Adverse Events (AEs) | From screening (day -28) until follow-up/early termination (ET) (Day 5 to Day 10 (after treatment Period 4/ET))
  To assess the adverse events as a criteria of safety and tolerability variables.
Vital sign (systolic and diastolic blood pressure [BP]) | At screening (Day -28), admission (Day -1), treatment periods 1, 2, 3, 4 (Day 1 - 3) and follow-up/ET (Day 5 to Day 10 (after treatment Period 4/ET))
  To assess the vital signs as a criteria of safety and tolerability variables.
Vital sign (pulse rate) | At screening (Day -28), admission (Day -1), treatment periods 1, 2, 3, 4 (Day 1 - 3) and follow-up/ET (Day 5 to Day 10 (after treatment Period 4/ET))
  To assess the vital signs as a criteria of safety and tolerability variables.
Twelve-lead electrocardiograms (ECGs) | At screening (Day -28) and follow-up/ET (Day 5 to Day 10 (after treatment Period 4/ET))
  To assess the cardiovascular system functioning as a criteria of safety and tolerability variables.
Physical examination | At screening (Day -28) and follow-up/ET (Day 5 to Day 10 (after treatment Period 4/ET))
  To assess the physical examination as a criteria of safety and tolerability variables.
Laboratory assessments (hematology and clinical chemistry) | At screening (Day -28), admission (day -1) and follow-up/ET (Day 5 to Day 10 (after treatment Period 4/ET))
  To assess the hematology and clinical chemistry as a criteria of safety and tolerability variables.
Laboratory assessments (Urinalysis (dipstick)) | At screening (Day -28), admission (day -1) and follow-up/ET (Day 5 to Day 10 (after treatment Period 4/ET))
  To assess the urinalysis as a criteria of safety and tolerability variables.

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Dr. med., Principal Investigator — PAREXEL Early Phase Clinical Unit Berlin
Locations (1):
- Research Site, Berlin, Germany

REFERENCES:
- [Derived] Niazi M, Wissmar J, Berggren AR, Karlsson C, Johanson P. Development Strategy and Relative Bioavailability of a Pediatric Tablet Formulation of Ticagrelor. Clin Drug Investig. 2019 Aug;39(8):765-773. doi: 10.1007/s40261-019-00800-w. PMID 31140114